CLINICAL TRIAL: NCT00475215
Title: A Multicenter, Randomized, Parallel Group, Comparative, Safety-Assessor Blinded, Phase IIIa Trial in Adult Surgical Subjects Under General Anesthesia at Increased Risk for Pulmonary Complications
Brief Title: Safety and Efficacy of Sugammadex (Org 25969, MK-8616) in Participants With or Having a Past History of Pulmonary Disease (19.4.308) (P05932) (MK-8616-017)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05932; 19.4.308 (Other: Organon Protocol Number); P05932 (Other: Schering-Plough Protocol Number); MK-8616-017 (Other: Merck Protocol Number)
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sugammadex; Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rocuronium + Sugammadex 2.0 mg/kg (Experimental): After the IV intubation dose (0.6 mg/kg) or last maintenance dose (0.15 mg/kg) of rocuronium, at reappearance of T2, participants will receive IV sugammadex 2.0 mg/kg.
  Interventions: Drug: Sugammadex; Drug: Rocuronium
- Rocuronium + Sugammadex 4.0 mg/kg (Experimental): After the IV intubation dose (0.6 mg/kg) or last maintenance dose (0.15 mg/kg) of rocuronium, at reappearance of T2, participants will receive IV sugammadex 4.0 mg/kg.
  Interventions: Drug: Sugammadex; Drug: Rocuronium

INTERVENTIONS:
Drug: Sugammadex — Sugammadex solution for injection.
  Other Names: Org 25969, MK-8616, Bridion®
Drug: Rocuronium — Rocuronium bromide solution for injection.
  Other Names: Zemuron®

SUMMARY:
The purpose of the trial is to research the safety and to show faster recovery after administration of 2.0 mg/kg or 4.0 mg/kg sugammadex (Org 25969, MK-8616) given as a reversal agent for 0.6 mg/kg (0.15 mg/kg maintenance dose) rocuronium (Zemuron®) in participants diagnosed with or having a history of pulmonary disease. All drug administration will be via the intravenous (IV) route.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class 1 to 3;
* Has been diagnosed with or having a past history of pulmonary disease;
* Is scheduled for elective surgical procedure under general anesthesia requiring neuromuscular block with the use of rocuronium;
* Is scheduled for surgery in supine position;
* Has given written informed consent;

Exclusion Criteria:

* Is expected to have a difficult intubation due to anatomical malformations;
* Has known or suspected of having neuromuscular disorders impairing neuromuscular blockade and/or significant renal dysfunction;
* Has known or suspected of having a (family) history of malignant hyperthermia;
* Has known or suspected of having an allergy to narcotics, muscle relaxants or other medications used during surgery;
* Is receiving medication known to interfere with neuromuscular blocking agents such as anticonvulsants, antibiotics and Mg2+;
* Is a female who is pregnant or breast-feeding;
* Is a female of childbearing potential not using an acceptable method of birth control [condom or diaphragm with spermicide, vasectomized partner (> 6 months), IUD, abstinence] or using only hormonal contraception as birth control;
* Has already participated in a sugammadex trial including Protocol 19.4.308;
* Has participated in another clinical trial, not pre-approved by Organon, within 30 days of entering into Protocol 19.4.308.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2005-10-27 (Actual); Primary Completion 2006-08-21 (Actual); Study Completion 2006-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Amao R, Zornow MH, Cowan RM, Cheng DC, Morte JB, Allard MW. Use of sugammadex in patients with a history of pulmonary disease. J Clin Anesth. 2012 Jun;24(4):289-97. doi: 10.1016/j.jclinane.2011.09.006. PMID 22608583
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 9 study sites in the United States.
Groups:
- Rocuronium + Sugammadex 2.0 mg/kg: After the intravenous (IV) intubation dose (0.6 mg/kg) or last maintenance dose (0.15 mg/kg) of rocuronium, at reappearance of T2, participants received IV sugammadex 2.0 mg/kg.
- Rocuronium + Sugammadex 4.0 mg/kg: After the IV intubation dose (0.6 mg/kg) or last maintenance dose (0.15 mg/kg) of rocuronium, at reappearance of T2, participants received IV sugammadex 4.0 mg/kg.
Period: Overall Study
Arm/Group | Rocuronium + Sugammadex 2.0 mg/kg | Rocuronium + Sugammadex 4.0 mg/kg
Started (Randomized) | 44 | 42
Treated | 39 | 38
Completed | 39 | 38
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Population: All treated participants are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rocuronium + Sugammadex 2.0 mg/kg | Rocuronium + Sugammadex 4.0 mg/kg | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49 (17) | 46 (14) | 47 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 57
  Male | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Time From Start of Sugammadex Administration to Recovery of T4/T1 Ratio to 0.9 in Participants With or Having a Past History of Pulmonary Disease
Description: The mean time from the start of sugammadex administration to recovery of the T4/T1 ratio to 0.9 was determined. Less time indicates faster recovery from neuromuscular blockade. The ratio of T4 (fourth twitch; amplitude of fourth response to train of four [TOF] stimulation is expressed as percent of control T4) over T1 (first twitch; amplitude of first response to TOF stimulation is expressed as percent of control T1) ranges from 0 (complete loss of T4 twitch response) to 1.0 (complete recovery of T4 twitch response). For TOF stimulation, 4 consecutive square wave supra-maximal stimuli of 0.2 msec duration were delivered at 2 Hz every 15 seconds. Neuromuscular monitoring was performed with the TOF-Watch® SX.
Time Frame: Up to 90 minutes
Population: All randomized participants who received sugammadex and had ≥1 post-baseline assessment of the outcome measure. For 11 participants (2.0 mg/kg n=6 and 4.0 mg/kg n=5), data were missing due to watch malfunction (n=2), the data that was obtained was considered unreliable (n=6), or the watch was removed prior to recovery to 0.9 (n=3).
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rocuronium + Sugammadex 2.0 mg/kg | Rocuronium + Sugammadex 4.0 mg/kg
Number analyzed (Participants) | 33 | 33
Minutes | 2.42 (1.93) | 2.1 (1.8)

2. Primary Outcome: Percentage of Participants Experiencing ≥1 Adverse Event(s) (AE)
Description: The percentage of participants experiencing ≥1 AE(s) was determined for each arm. An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: Up to 7 days
Population: All randomized participants who received sugammadex are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Rocuronium + Sugammadex 2.0 mg/kg | Rocuronium + Sugammadex 4.0 mg/kg
Number analyzed (Participants) | 39 | 38
Percentage of Participants | 97.4 | 94.7

3. Primary Outcome: Percentage of Participants Discontinuing Study Treatment Due to an Adverse Event (AE)
Description: The percentage of participants discontinuing from study treatment due to an AE was determined for each arm. An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: Up to 7 days
Population: All randomized participants who received sugammadex are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Rocuronium + Sugammadex 2.0 mg/kg | Rocuronium + Sugammadex 4.0 mg/kg
Number analyzed (Participants) | 39 | 38
Percentage of Participants | 0 | 0

4. Secondary Outcome: Time From Start of Sugammadex Administration to Recovery of T4/T1 Ratio to 0.7 in Participants With or Having a Past History of Pulmonary Disease
Description: The mean time from the start of sugammadex administration to recovery of the T4/T1 ratio to 0.7 was determined. Less time indicates faster recovery from neuromuscular blockade. The ratio of T4 (fourth twitch; amplitude of fourth response to train of four [TOF] stimulation is expressed as percent of control T4) over T1 (first twitch; amplitude of first response to TOF stimulation is expressed as percent of control T1) ranges from 0 (complete loss of T4 twitch response) to 1.0 (complete recovery of T4 twitch response). For TOF stimulation, 4 consecutive square wave supra-maximal stimuli of 0.2 msec duration were delivered at 2 Hz every 15 seconds. Neuromuscular monitoring was performed with the TOF-Watch® SX.
Time Frame: Up to 90 minutes
Population: All randomized participants who received sugammadex and had ≥1 post-baseline assessment of the outcome measure. For 6 participants (2.0 mg/kg n=3 and 4.0 mg/kg n=3), data were unavailable due to TOF-Watch® malfunction (n=2), or the data that was obtained was considered unreliable (n=4).
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rocuronium + Sugammadex 2.0 mg/kg | Rocuronium + Sugammadex 4.0 mg/kg
Number analyzed (Participants) | 36 | 35
Minutes | 1.5 (0.55) | 1.35 (0.45)

5. Secondary Outcome: Time From Start of Sugammadex Administration to Recovery of T4/T1 Ratio to 0.8 in Participants With or Having a Past History of Pulmonary Disease
Description: The mean time from the start of sugammadex administration to recovery of the T4/T1 ratio to 0.8 was determined. Less time indicates faster recovery from neuromuscular blockade. The ratio of T4 (fourth twitch; amplitude of fourth response to train of four [TOF] stimulation is expressed as percent of control T4) over T1 (first twitch; amplitude of first response to TOF stimulation is expressed as percent of control T1) ranges from 0 (complete loss of T4 twitch response) to 1.0 (complete recovery of T4 twitch response). For TOF stimulation, 4 consecutive square wave supra-maximal stimuli of 0.2 msec duration were delivered at 2 Hz every 15 seconds. Neuromuscular monitoring was performed with the TOF-Watch® SX.
Time Frame: Up to 90 minutes
Population: All randomized participants who received sugammadex and had ≥1 post-baseline assessment of the outcome measure. For 7 participants (2.0 mg/kg n=4 and 4.0 mg/kg n=3), data were unavailable due to TOF-Watch® malfunction (n=2), or the data that was obtained was considered unreliable (n=5).
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rocuronium + Sugammadex 2.0 mg/kg | Rocuronium + Sugammadex 4.0 mg/kg
Number analyzed (Participants) | 35 | 35
Minutes | 1.8 (0.82) | 1.62 (0.65)

6. Secondary Outcome: Level of Consciousness Assessment 1: Prior to Transfer to the Recovery Room Following Extubation
Description: The level of consciousness prior to transfer to the recovery room was determined by the clinician for each participant. Each participants was assigned 1 of 3 potential levels of consciousness: 1) awake and oriented; 2) arousable with minimal stimulation; or 3) responsive only to tactile stimulation.
Time Frame: Up to 6 hours (prior to transfer to the recovery room after extubation)
Population: All randomized participants who received sugammadex and had ≥1 post-baseline assessment for the outcome measure. One participant in the 4.0 mg/kg group had missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium + Sugammadex 2.0 mg/kg | Rocuronium + Sugammadex 4.0 mg/kg
Number analyzed (Participants) | 39 | 38
Participants
  Awake and oriented | 17 | 22
  Arousable with minimal stimulation | 16 | 13
  Responsive only to tactile stimulation | 6 | 2
  Missing data | 0 | 1

7. Secondary Outcome: Level of Consciousness Assessment 2: Prior to Discharge From the Recovery Room
Description: The level of consciousness prior to discharge from the recovery room was determined by the clinician for each participant. Each participants was assigned 1 of 3 potential levels of consciousness: 1) awake and oriented; 2) arousable with minimal stimulation; or 3) responsive only to tactile stimulation.
Time Frame: Up to 6 hours (prior to discharge from the recovery room)
Population: All randomized participants who received sugammadex and had ≥1 post-baseline assessment for the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium + Sugammadex 2.0 mg/kg | Rocuronium + Sugammadex 4.0 mg/kg
Number analyzed (Participants) | 39 | 38
Participants
  Awake and oriented | 38 | 38
  Arousable with minimal stimulation | 1 | 0
  Responsive only to tactile stimulation | 0 | 0

8. Secondary Outcome: Five-Second Head Lift Assessment 1: Prior to Transfer to the Recovery Room Following Extubation
Description: The ability of each cooperative (based on clinician determination) participant to perform a 5-second head lift was determined by the clinician. Participants were rated as either able or not able to complete the head lift task.
Time Frame: Up to 6 hours (prior to transfer to the recovery room after extubation)
Population: All randomized and cooperative participants who received sugammadex and had ≥1 post-baseline assessment of the outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium + Sugammadex 2.0 mg/kg | Rocuronium + Sugammadex 4.0 mg/kg
Number analyzed (Participants) | 28 | 34
Participants
  Able to perform | 23 | 29
  Not able to perform | 5 | 5

9. Secondary Outcome: Five-Second Head Lift Assessment 2: Prior to Discharge From the Recovery Room
Description: as for outcome 8
Time Frame: Up to 6 hours (prior to discharge from the recovery room)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium + Sugammadex 2.0 mg/kg | Rocuronium + Sugammadex 4.0 mg/kg
Number analyzed (Participants) | 39 | 38
Participants
  Able to perform | 39 | 37
  Not able to perform | 0 | 1

10. Secondary Outcome: General Muscle Weakness Assessment 1: Prior to Transfer to the Recovery Room Following Extubation
Description: Each cooperative (based on clinician determination) participant was assessed by a clinician to determine if there was muscle weakness. Participants were rated as having or not having muscle weakness by the clinician.
Time Frame: Up to 6 hours (prior to transfer to the recovery room after extubation)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium + Sugammadex 2.0 mg/kg | Rocuronium + Sugammadex 4.0 mg/kg
Number analyzed (Participants) | 28 | 34
Participants
  Muscle Weakness | 3 | 4
  No Muscle Weakness | 25 | 30

11. Secondary Outcome: General Muscle Weakness Assessment 2: Prior to Discharge From the Recovery Room
Description: as for outcome 10
Time Frame: Up to 6 hours (prior to discharge from the recovery room)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Rocuronium + Sugammadex 2.0 mg/kg | Rocuronium + Sugammadex 4.0 mg/kg
Number analyzed (Participants) | 39 | 38
Participants
  Muscle Weakness | 4 | 6
  No Muscle Weakness | 35 | 32

ADVERSE EVENTS:
Time Frame: Up to 7 days
Description: All randomized participants who received sugammadex are included.
Groups:
- Rocuronium + Sugammadex 2.0 mg: After the IV intubation dose (0.6 mg/kg) or last maintenance dose (0.15 mg/kg) of rocuronium, at reappearance of T2, participants received IV sugammadex 2.0 mg/kg.
- Rocuronium + Sugammadex 4.0 mg: After the IV intubation dose (0.6 mg/kg) or last maintenance dose (0.15 mg/kg) of rocuronium, at reappearance of T2, participants received IV sugammadex 4.0 mg/kg.
Arm/Group | Rocuronium + Sugammadex 2.0 mg | Rocuronium + Sugammadex 4.0 mg
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/38
Serious Adverse Events (participants affected / at risk) | 4/39 | 3/38
Other Adverse Events (participants affected / at risk) | 38/39 | 34/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocuronium + Sugammadex 2.0 mg (N=39) | Rocuronium + Sugammadex 4.0 mg (N=38)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Poor peripheral circulation (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocuronium + Sugammadex 2.0 mg (N=39) | Rocuronium + Sugammadex 4.0 mg (N=38)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Flatulence (Gastrointestinal disorders) | 4 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 13 (19) | 9 (10)
Vomiting (Gastrointestinal disorders) | 7 (7) | 5 (5)
Chills (General disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 2 (2)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Incision site complication (Injury, poisoning and procedural complications) | 8 (16) | 7 (8)
Incision site haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Post procedural nausea (Injury, poisoning and procedural complications) | 3 (3) | 4 (6)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Procedural hypertension (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Procedural hypotension (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 27 (28) | 27 (30)
Beta 2 microglobulin increased (Investigations) | 2 (2) | 0 (0)
Haemoglobin decreased (Investigations) | 5 (5) | 1 (1)
Urine output decreased (Investigations) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any such scientific paper, presentation, or other communication concerning the clinical trial described in this protocol will first be submitted to the Sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.